CLINICAL TRIAL: NCT06782685
Title: Liposomal Irinotecan in Combination With Oxaliplatin and Bevacizumab Versus Liposomal Irinotecan in Combination With 5-FU/LV for the Second-line Treatment of Advanced Pancreatic Cancer
Brief Title: Liposomal Irinotecan + Oxaliplatin + Bevacizumab Versus Liposomal Irinotecan + 5-FU/LV
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dai, Guanghai (Other)
Responsible Party: Sponsor-Investigator, Dai, Guanghai, chief physician, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DNY-PC-B01
Record Dates: First submitted 2024-10-10; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Advanced Pancreatic Cancer (Part 1)
MeSH Terms: interventions — Oxaliplatin; Bevacizumab; Fluorouracil; irinotecan sucrosofate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Irinotecan liposomal combination of oxaliplatin and bevacizumab (Experimental): To explore the optimal dose combination of irinotecan liposomes plus oxaliplatin in the regimen of irinotecan liposomes plus oxaliplatin in bevacizumab and determine the recommended dose for phase II
  Interventions: Drug: Irinotecan liposoma; Drug: oxaliplatin; Drug: bevacizumab
- Irinotecan liposomal combination of 5-FU/LV (Active Comparator): Standard treatment
  Interventions: Drug: 5-FU; Drug: LV; Drug: Irinotecan Liposomal
- Irinotecan liposomal +oxaliplatin +bevacizumab (Experimental): Phase II recommended dose
  Interventions: Drug: bevacizumab; Drug: Irinotecan Liposomal; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Irinotecan liposoma — Exploration started with 50mg/m^2 dose, preset 50mg/m^2, 60mg/m^2, 2 dose groups, IV infusion 90min, d1
  Arms: Irinotecan liposomal combination of oxaliplatin and bevacizumab
Drug: oxaliplatin — Exploration started with 60mg/m^2 dose, preset 60mg/m^2, 85mg/m^2, 2 dose groups, IV infusion, d1
  Arms: Irinotecan liposomal combination of oxaliplatin and bevacizumab
Drug: bevacizumab — 5mg/kg，i.v.，d1
  Arms: Irinotecan liposomal +oxaliplatin +bevacizumab; Irinotecan liposomal combination of oxaliplatin and bevacizumab
Drug: 5-FU — 2400mg/m^2, i.v.，46h
  Arms: Irinotecan liposomal combination of 5-FU/LV
Drug: LV — 400mg/m^2, i.v.，d1
  Arms: Irinotecan liposomal combination of 5-FU/LV
Drug: Irinotecan Liposomal — 70mg/m^2, i.v.，d1
  Arms: Irinotecan liposomal combination of 5-FU/LV
Drug: Irinotecan Liposomal — Phase II recommended dose
  Arms: Irinotecan liposomal +oxaliplatin +bevacizumab
Drug: Oxaliplatin — Phase II recommended dose
  Arms: Irinotecan liposomal +oxaliplatin +bevacizumab

SUMMARY:
Purpose of the study Phase I study: to explore the optimal dose combination of irinotecan liposome + oxaliplatin + bevacizumab regimen, irinotecan liposome + oxaliplatin Phase II study: to evaluate the safety and efficacy of the second-line treatment regimen of irinotecan liposome combined with oxaliplatin and bevacizumab compared to the second-line treatment regimen of irinotecan liposome combined with 5-FU/LV in advanced pancreatic cancer Sample size 138 cases Phase I Crawl, sample size 9-18 cases. Phase II randomized controlled clinical study, historical data NAPOLI-1 study, ORR of 8.8% for irinotecan liposome + 5-FU/LV, planned trial arm ORR upgrade to 25%, calculated at 60 cases in each arm.

Subject population Patients with advanced pancreatic cancer diagnosed after failure of first-line therapy, confirmed by histopathology or cytopathology, who meet the inclusion criteria and do not meet the exclusion criteria.

Phase I design:

Liposomal irinotecan + oxaliplatin + bevacizumab, 2-week regimen Liposomal irinotecan: start exploring with 50mg/m2 dose, preset 50mg/m2, 60mg/m2, 2 dose groups, 90min IV infusion, d1; Oxaliplatin: explored from 60mg/m2 dose, preset 60mg/m2, 85mg/m2, 2 dose groups, IV infusion, d1; Bevacizumab: 5 mg/kg, i.v., d1; Phase II study design.

Trial group:

Irinotecan liposomal: RP2D, i.v., 90min, d1; Oxaliplatin: RP2D, i.v., d1; Bevacizumab: 5mg/kg, i.v., d1; Cycles every 2 weeks until disease progression or intolerable; imaging every 3 treatment cycles/1.5 months.

Control:

Liposomal irinotecan: 70 mg/m2 IV for 90 min, d1; Calcium folinate: 400 mg/m2, IV infusion over 30 min, d1; 5-FU: 2400 mg/m2, continuous IV infusion over 46h; Cycles every 2 weeks until disease progression or intolerable; imaging every 3 treatment cycles/1.5 months.

Notes:

If the duration of irinotecan liposome infusion can be extended appropriately based on the patient's clinical response; if the patient withdraws from the trial due to intolerance of toxicity (e.g., neurotoxicity or myelotoxicity) induced by one of the drugs, follow up is required until PFS and OS.

Translated with DeepL.com (free version)

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years old;
2. Patients with pancreatic cancer diagnosed by histopathology or cytology;
3. Unresectable disease assessed by multidisciplinary and imaging;
4. Subjects who have received prior failed first-line therapy, and recurrence within 6 months of the end of (neo)adjuvant therapy is considered a first-line treatment failure;
5. Subjects who have not received platinum-containing or irinotecan drugs for prior first-line therapy;
6. Patients with at least one evaluable lesion according to RECIST v1.1;
7. ECOG score of 0-2;
8. Expected survival ≥ 3 months;
9. Bone marrow function: absolute neutrophil count (ANC) ≥1.5×10^9/L, hemoglobin ≥90 g/dL, platelets (PLT) ≥100×10^9/L, and white blood cells (WBC) ≥3.0×10^9/L;
10. Liver function: alanine aminotransferase (ALT), alanine aminotransferase (AST), alkaline phosphatase (ALP) ≤2.5 times the upper limit of normal (ULN), or ≤5×ULN if liver metastases are present, total bilirubin<1.5 ULN;
11. Renal function: serum creatinine (Cr) ≤1.5 × ULN or creatinine clearance (CCr) ≥60 mL/min (according to the Cockcroft-Gault formula);
12. Coagulation function: prothrombin time (PT), activated partial thromboplastin time (APTT) and international normalized ratio (INR) ≤1.5 × ULN;
13. Patients with biliary obstruction should receive adequate biliary drainage; and
14. Adverse reactions arising from prior therapy must be restored to grade 1 or baseline according to CTCAE 5.0 (with the exception of toxicities such as alopecia, grade 2 or lower peripheral neuropathy, which can be enrolled with no safety risk in the judgment of the investigator);
15. Non-pregnant or lactating females; females/males of childbearing potential should use effective contraception during the study and for 6 months after completion of study treatment;
16. Patients are compliant, understand the study procedures, and sign a written informed consent form.

Exclusion Criteria:

1. Patients who have had other malignant tumors within the previous 5 years (except cured carcinoma in situ and basal cell carcinoma of the skin);
2. Uncontrollable pleural effusion or ascites;
3. Any known brain metastasis or meningeal metastasis;
4. Concomitant use of a potent CYP3A4 inducer within 3 weeks prior to the first dose, or concurrent use of a potent CYP3A4 inhibitor or potent UGT1A1 inhibitor within 3 weeks prior to the first dose;
5. Patients undergoing major organ surgery (except needle biopsy, central venous catheterization, port catheterization, stent placement for relief of biliary obstruction, percutaneous hepato-biliary drainage, cholecystostomy) or elective surgical procedures scheduled within 4 weeks prior to the first dose of study drug;
6. Systemically treated active, uncontrolled bacterial, viral, or fungal infections, defined as persistent signs/symptoms associated with the infection that do not improve despite appropriate antibiotics, antiviral therapy, and/or other treatments;
7. Subjects with congenital or acquired immunodeficiency, such as HIV-infected individuals or active hepatitis (transaminases do not meet the inclusion criteria, Hepatitis B : HBV DNA ≥ 1000 IU/ml; Hepatitis C : HCV RNA ≥ 1000 IU/ml); chronic hepatitis B viral carriers, with HBV DNA < 2000 IU/ml, who must be concurrently receiving antiviral during the trial period treatment before enrollment;
8. Presence of serious concomitant diseases: those with diabetes mellitus that cannot be well controlled by glucose-lowering drugs, difficult-to-control hypertension, severe cardiovascular and cerebral vascular disease, renal failure, hepatic failure, uncontrolled epilepsy, central nervous system disease or history of mental disorders, those with a clear tendency to gastrointestinal bleeding, intestinal paralysis, intestinal obstruction, etc;
9. >grade 1 diarrhea with an increase in the number of bowel movements >4 times per day compared to baseline; moderate to severe increase in stoma discharge; limited instrumental activities of daily living or even limited spontaneous activities of daily living; life-threatening; requiring urgent treatment;
10. Those with serum albumin ≤ 3 g/dL;
11. Those who had participated in other clinical studies within 4 weeks prior to enrollment;
12. Patients assessed by the investigator to be unsuitable for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2024-06-23 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
To explore the optimal dose combination of irinotecan liposomes plus oxaliplatin in the regimen of irinotecan liposomes plus oxaliplatin in bevacizumab | At the end of Cycle 1 (each cycle is 14 days)
  The DLT determination criteria are as follows:
  1. Hematologic toxicity：
     * Grade 4 neutropenia with application of granulocyte colony-stimulating factor still persisting for >3 days ;
     * Grade 3 or above FN;
     * Grade 3 thrombocytopenia with bleeding and/or need for blood transfusion;
     * Grade 4 thrombocytopenia;
     * Grade 4 anemia.
  2. Non-hematologic toxicity： ≥ Grade 3 non-hematologic toxicity, except: ① Transient (≤24 hours) Grade 3 fever (>40°C), Grade 3 malaise, Grade 3 headache, Grade 3 nausea, which recovers to Grade 1 or baseline after treatment; Grade 3 vomiting, Grade 3 electrolyte disorders (including hypokalemia, hypophosphatemia, hypocalcemia, etc.), recovery to Grade 1 or baseline within 48 hours after treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing, Beijing
  - Chinese PLA General Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://gco.iarc.fr/today/data/factsheets/cancers/13-Pancreas-fact-sheet.